CLINICAL TRIAL: NCT03195361
Title: Multicenter, Prospective, Non-randomized, Single-arm, Interventional Study for the Evaluation of the Safety and Preformance of the SRS Device for the Treatment of Pelvic Organ Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lyra Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-14-011
Record Dates: First submitted 2016-05-01; First posted 2017-06-22 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Anterior Vaginal Wall Prolapse With/Without Apical/Uterine Descent

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm (Experimental): Subjects suffering from anterior POP-Q grade 2 (point Aa and Ba≥ -1) and above, who are scheduled for POP surgery, will be transplanted with the SRS device
  Interventions: Device: SRS - Self Retaining Support system

INTERVENTIONS:
Device: SRS - Self Retaining Support system
  Other Names: transvaginal surgical treatment

SUMMARY:
A prospective, single arm, multi-center clinical study to evaluate the safety and performance of the SRS (Lyra Medical) vaginal mesh in POP patients

DETAILED DESCRIPTION:
The SRS implant is intended for transvaginal surgical treatment of anterior vaginal wall prolapse with or without vaginal apex/uterine prolapses

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed the informed consent form and is willing to participate in the clinical study and data collection.
2. Patient age is between 50 and 75 years old
3. POP-Q: Aa and/or Ba is at least -1

Exclusion Criteria:

1. Patient is pregnant or breastfeeding
2. Patient is suffering from active infection (on antibiotic therapy)
3. Patient is planning vaginal delivery
4. Patient had previous vaginal mesh surgery
5. Patient is in high risk for surgery (evidence of clinically significant cardiovascular, renal, hepatic, coagulatory or respiratory diseases).
6. Any condition that in the judgment of the investigators would interfere with the subject's ability to provide informed consent, comply with study instructions, place the subject at increased risk, or which might confound interpretation of study results.
7. Malignancy.
8. Known hypersensitivity to PEEK and/or polypropylene materials.
9. Participation in another investigational trial that has not completed the primary endpoint or interferes with study participation.
10. Diagnosed with mental or emotional disturbance.

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Improvement in POP-Q points Aa and Ba | 36 months
  Points Aa and\or Ba are less than -1
Improvement in POP-Q point C: | 36 months
  Point C at -5 or less
No unexpected serious adverse device related events | 36 months

SECONDARY OUTCOMES:
Achieving normal urinary function: | 36 Months
  Patient does not experience voiding dysfunction and have negative Urinary Cough Test.
Improvement in Quality Of Life (QoL) | 36 Months
  Subjective bother involving pelvic floor disorders using validated scales including PFDI-20 and PSIQ-12.

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Mayanei HaYeshua Medical Center, Bnei Brak
  - Ziv Medical center, Safed
  - Asaf HaRofeh Medical Center, Zrifin